CLINICAL TRIAL: NCT00376428
Title: Application of Functional Electrophysiological Tests to Evaluate Pharmacological Treatments in Patients With Cystic Fibrosis
Brief Title: Interest of Gentamicin-induced Readthrough in Cystic Fibrosis Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-03-10
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2006-09

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis Transmembrane Conductance Regulator; Premature termination codon; Gentamicin-induced readthrough
MeSH Terms: conditions — Cystic Fibrosis | interventions — Gentamicins

INTERVENTIONS:
Drug: Gentamicin

SUMMARY:
Suppression of stop mutations in the CFTR gene with parenteral gentamicin can be predicted in vitro and is associated with clinical benefit and significant modification of the CFTR-mediated chloride transport in nasal and sweat gland epithelium.

DETAILED DESCRIPTION:
Background: This study was conducted to determine whether intravenous gentamicin can suppress stop codons in cystic fibrosis (CF) patients and, if so, whether it has any clinical benefits.

Methods: We first used a dual gene reporter system to determine the gentamicin-induced readthrough level of the most frequent CFTR stop mutations in the French population. We next investigated readthrough efficiency in response to 10 mg/kg once daily intravenous gentamicin perfusions in patients with stop mutations and in a control group of patients without stop mutations. Respiratory function, sweat chloride concentration, nasal potential difference (NPD) and CFTR expression in nasal epithelial cells were measured at baseline and after 15 days of treatment.

Results: After in vitro gentamicin incubation, the readthrough efficiency for the Y122X mutation was at least five times higher than that for G542X, R1162X, and W1282X. In six of the nine patients with the Y122X mutation, CFTR immunodetection showed protein expression at the membrane of the nasal ciliated cells and the CFTR-dependent chloride secretion in their NPD measurements increased significantly. Respiratory status also improved in these patients, irrespective of the gentamicin sensitivity of the germs present in the sputum. Mean sweat chloride concentration decreased significantly and normalized in two patients. These measurements did not change in the Y122X patients with no protein expression, in patients with the other stop mutations investigated in vitro (n=4) and those without stop mutations (n=5).

Conclusion: Suppression of stop mutations in the CFTR gene with parenteral gentamicin can be predicted in vitro and is associated with clinical benefit and significant modification of the CFTR-mediated chloride transport in nasal and sweat gland epithelium.

ELIGIBILITY:
Inclusion Criteria:

* cystic fibrosis with CFTR codon stop mutations

Exclusion Criteria:

* Rhinitis
* nasal polyposis
* passive or active smoking
* modification of basal treatments within the previous month
* treatments with aminoglycosides within three previous months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2003-01; Study Completion 2005-06

PRIMARY OUTCOMES:
CFTR-dependant chlorate secretion

SECONDARY OUTCOMES:
CFTR expression in nasal cells
Clinical beneficial effects

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Edelman, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France; Isabelle Sermet, MD; PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker-Enfants malades, Paris, France